CLINICAL TRIAL: NCT07281118
Title: Intercostal Cryoanalgesia in Double Lung Transplant Recipients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: AtriCure, Inc. (Industry)
Responsible Party: Principal Investigator, Abbas Ardehali, MD, Professor of Surgery and Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-24-6029
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Post-operative Pain Management
Keywords: Lung Transplant; Pain Management
MeSH Terms: conditions — Agnosia | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Patients will be treated intra-operatively with Atricure CryoSPHERE MAX Probe to 2
  Interventions: Device: Atricure CryoSPHERE MAX Probe
- Usual Care (No Intervention): No treatment intra-operatively

INTERVENTIONS:
Device: Atricure CryoSPHERE MAX Probe — Patients will be treated intra-operatively with Atricure CryoSPHERE MAX Probe to 2 intercostal spaces above and below the thoracotomy incision for 1 minutes for each application during their double lung transplant procedure.
  Other Names: Cryotherapy
  Arms: Treatment Arm

SUMMARY:
This study is testing a new way to help manage pain after a double lung transplant. Instead of relying only on strong pain medicines like opioids, doctors will use a cold-therapy probe during surgery to help numb the nerves near the incision. Researchers want to see if this method can reduce the need for opioids and improve recovery.

DETAILED DESCRIPTION:
This study is being done to learn whether a special cold-therapy treatment can help control pain after a double lung transplant. During the surgery, doctors may use a device called the Atricure CryoSPHERE MAX Probe, which gently freezes the nerves around the incision to reduce pain for several days. This freezing effect may help patients need fewer opioid pain medicines, which can sometimes cause sleepiness or make it harder to breathe deeply after surgery. Researchers will compare patients who receive the cryotherapy treatment to patients who receive the usual care without the device.

The main goal is to see whether the cryotherapy group uses at least 25% fewer opioids in the first 10 days after surgery. The study will also look at how often patients still need extra pain treatments, such as an epidural, and whether their average daily pain scores are lower. Another important question is whether the treatment can help shorten the amount of time patients need to stay in the ICU. About 148 people from several hospitals will take part in the study. Everyone who joins the study will be followed for one year after their transplant to monitor their recovery and any long-term effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Undergoing double lung transplantation via bilateral thoracotomies or clamshell incision

Exclusion Criteria:

* Multi-organ transplant recipients
* Redo lung transplant recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-11-24 (Estimated); Study Completion 2027-11-24 (Estimated)

PRIMARY OUTCOMES:
Total opioid use (oral morphine equivalents) | 1 year
  Total opioid use (oral morphine equivalents)

SECONDARY OUTCOMES:
Frequency of rescue therapy | 1 year
  Compare need for thoracic epidural anesthesia.
Median daily pain score | Day 10
  To compare the Median daily pain score for the first 10 days after lung transplantation, Numerical Rating Scale (NRS) (0-10): A standard 11-point scale (0=no pain, 10=worst imaginable pain) used for pain intensity, showing good reliability and validity in various conditions like neuropathic pain.
Duration of ICU Stay | Days 1-10, 30 days, 60 days
  To compare the duration of the ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Ardehali, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Baylor University, Waco, Texas

IPD SHARING:
Plan to Share IPD: No
Summary data and results will be shared.